CLINICAL TRIAL: NCT04979156
Title: LaserEn: SOLTIVE™ Thulium Laser Fiber En Bloc Resection of Bladder Tumors
Acronym: LaserEn
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Holzbeierlein, Principal Investigator, University of Kansas Medical Center
Other Study IDs: LaserEn
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer; Surgery
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SOLTIVE™ Thulium Laser Fiber En Bloc Resection of Bladder Tumors: SOLTIVE™ Thulium Laser Fiber En Bloc Resection of Bladder Tumors
  Interventions: Procedure: SOLTIVE™ Thulium Laser Fiber En Bloc Resection of Bladder Tumors

INTERVENTIONS:
Procedure: SOLTIVE™ Thulium Laser Fiber En Bloc Resection of Bladder Tumors — SOLTIVE™ Thulium Laser Fiber En Bloc Resection of Bladder Tumors
  Other Names: TURBT En Bloc

SUMMARY:
Conventional monopolar or bipolar transurethral resection of bladder tumors is the most common method for resection of a bladder mass. En bloc resection has demonstrated success in the literature utilizing different techniques and lasers, including utilizing the Ho:YAG and Tm:YAG lasers. A recent metanalysis revealed several benefits to laser en bloc resection including less complications and lower recurrence rate.22 Subsequently, laser technology has also advanced with the development of a super pulsed TFL which overcomes many limitations of prior traditional lasers. Olympus' SOLTIVE™ TFL, which has demonstrated improved maneuverability and control, has a shallow depth of tissue penetration at 0.15mm leading to precise resection and optimal hemostasis. Despite these beneficial characteristics and qualities along with the promising utility of en bloc resection, the Olympus SOLTIVE™ TFL has not been described in en bloc resection of bladder tumors. The investigator seek to determine if the proposed benefits of this device can be realized both pathologically and clinically in en bloc resection of bladder tumors.

DETAILED DESCRIPTION:
This is a prospective study investigating the use of the SOLTIVE™ Thulium Super pulse laser for the treatment of bladder tumors via en bloc resection in patients who present for treatment at the University of Kansas Health System. The study pretreatment evaluation and follow up schedule are the same as used routinely in daily practice, in accordance with standard of care practices. Routine labs (e.g. complete blood count, basic or complete metabolic panel, urinalysis and urine culture), and imaging will be obtained as per standard care at the provider's discretion based on the patient's history and physical exam.

A prospective data collection of the patients with bladder cancer undergoing en bloc resection will be conducted in this study.

A complete medical, surgical and bladder cancer history will be obtained by the surgical team in the pre-operative setting, per standard of care practices.

Patients will be taken to the operating room per standard of care for resection of one or more bladder tumors. The SOLTIVE™ Super Pulsed Thulium laser will be utilized for resection of the tumors in an en bloc fashion.

Technique for en bloc resection of bladder tumor Tumor marked with a circular coagulation blockage border approximately 1.0 cm away from the edge. All visible vessels around the tumor will be coagulated and lasered before the incision to reduce bleeding. Along this mark, a fan-shaped incision into the bladder wall is made until the muscle layer is visible uplift tumor by the force of the irrigation and use of the laser tip, gradually exposing the tumor base tumor base is disconnected tumor is then removed en bloc. If it is unable to be removed through the resectoscope in one piece due to its size, it may be cut into 2 pieces at the surgeon's discretion.

At the surgeon's discretion, the procedure may be converted to a traditional TURBT utilizing either monopolar or bipolar loop electrocautery. Other intraoperative/postoperative decisions based on surgeon discretion and standard of care treatment:

Each specimen will be collected and sent en bloc to the pathology department. Ameer Hazma, MD, a genitourinary pathologist, will review all specimens to decrease interobserver variation.

Urinary symptoms before and after the procedure will be evaluated. This will be assessed via an electronic questionnaire that will be sent to study participants. Symptoms will be evaluated pre-operatively the morning of surgery as well as on post-operative day #3, 7, and 14.

No validated questionnaire for evaluation of urinary symptoms after bladder tumor resection currently exists. From clinical experience, the symptoms patients most commonly report include frequency, urgency, dysuria, or hematuria. The investigator will therefore modified the existing American Urological Association's Symptom score to address these symptoms on a shorter term basis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patient presenting for resection of papillary bladder tumor visualized on cystoscopy

   1. New bladder tumor
   2. Recurrent tumors
3. Tumor <3cm

Exclusion Criteria:

1. Patient unwilling to undergo en bloc resection
2. Non papillary lesions/tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing resection of the bladder for bladder tumors.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the ability to obtain identifiable pathologic characteristics of bladder tumor specimens by use the SOLTIVE™ laser during en bloc resection. | 6 months
  To determine the ability to obtain identifiable pathologic characteristics of bladder tumor specimens by use the SOLTIVE™ laser during en bloc resection.

SECONDARY OUTCOMES:
To evaluate the overall recurrence rate as well as the recurrence rate at the prior resection site after SOLTIVE™ en bloc resection of bladder tumors. | 6 months
  To evaluate the overall recurrence rate as well as the recurrence rate at the prior resection site after SOLTIVE™ en bloc resection of bladder tumors.
To evaluate patient symptoms before and after en bloc tumor resection | 6 months
  To evaluate patient symptoms before and after en bloc tumor resection
• To evaluate short-term complications within 3 months after SOLTIVE™ en bloc resection of bladder tumors. | 6 months
  • To evaluate short-term complications within 3 months after SOLTIVE™ en bloc resection of bladder tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Holzbeierlein, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No